CLINICAL TRIAL: NCT00508950
Title: Blood Collection In Healthy Adult Volunteers To Obtain Serum For Use In Pneumococcal Opsonophagocytic Assay Development.
Brief Title: Study Evaluating Serum Collected From Healthy Adults For Development of Pneumococcal Opsonophagocytic Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group
Other Study IDs: 6115A1-1000; B1851075 (Other: Alias Study Number)
Record Dates: First submitted 2007-07-27; First posted 2007-07-30 (Estimated); Last update posted 2016-08-17 (Estimated); Status verified 2016-08

CONDITIONS: Healthy
Keywords: Vaccines; Pneumococcal Conjugate Vaccine; Adult

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All subjects (Other): All subjects
  Interventions: Procedure: Large volume blood draw

INTERVENTIONS:
Procedure: Large volume blood draw — Large volume blood draw

SUMMARY:
The study will identify healthy adults who have been vaccinated against pneumococcus, and collect blood for the purpose of developing laboratory assays.

DETAILED DESCRIPTION:
Collect serum with antibody levels capable of killing pneumococcal bacteria from healthy prevaccinated adults to develop OPA assays for the 13 serotypes in 13-valent pneumococcal conjugate vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults 18-70 years of age
* Must have received 23vPS pneumococcal vaccine

Exclusion Criteria:

* Bleeding diathesis
* Pregnancy
* Chronic disease which could be worsened by donating blood
* Receipt of blood, blood products or immune globulin within six months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 152 (Actual)
Dates: Start 2007-08; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
To identify potential serum donors and obtain unit volumes of blood from these donors for use in pneumococcal opsonophagocytic assay development. | 8 years

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Frontage Clinical Services Inc., Secaucus, New Jersey, United States

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=6115A1-1000&StudyName=Study%20Evaluating%20Serum%20Collected%20From%20Healthy%20Adults%20For%20Development%20of%20Pneumococcal%20Opsonophagocytic%20Assay